CLINICAL TRIAL: NCT07099313
Title: Association of Prophylactic Treatment With Treatment Burden, Self-efficacy, Adherence, Sleep Quality, and Locus of Control in Patients With Hemophilia; an Ambispective Cohort Study
Brief Title: Association of Prophylactic Treatment With Treatment Burden and Psychosocial Variables in Patients With Hemophilia
Status: Recruiting | Type: Observational
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, Principal Investigator, Investigación en Hemofilia y Fisioterapia
Other Study IDs: He-ProF
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia
Keywords: Hemophilia; Clotting factor concentrates; Treatment burden; Perceived self-efficacy; Adherence; Locus of control
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients diagnosed with hemophilia A or B, undergoing prophylactic treatment with short half-life (SHL) and extended half-life (EHL) clotting factor concentrates.

SUMMARY:
Introduction: Hemophilia is a congenital coagulopathy characterised by recurrent haemarthrosis, leading to chronic arthropathy and functional impairment. Prophylactic treatment with extended half-life (EHL) or short half-life (SHL) clotting factor concentrates is the most effective strategy for preventing these episodes. EHL products have demonstrated haemostatic efficacy, with a lower frequency of infusions, potentially reducing the treatment burden, although their psychosocial impact has not yet been sufficiently explored.

Objectives: To evaluate the association between perceived treatment burden and psychosocial variables such as self-efficacy, adherence, sleep quality and health locus of control, depending on the type of treatment received (EHL or SHL).

Methods. Multicentre, ambispective cohort study. A total of 114 patients with haemophilia A or B undergoing EHL or SHL prophylactic treatment will be included. The primary variable will be treatment burden (Treatment Burden Questionnaire). Secondary variables will be perceived self-efficacy (General Self-Efficacy Scale), adherence (Torres scale), sleep quality (Pittsburgh Sleep Quality Index), treatment adherence (Torres Questionnaire) and health locus of control (Multidimensional Health Locus of Control). Potential confounding variables will include sociodemographic data (age, educational level, living arrangements) and clinical data (number of weekly infusions, type of hospital).

Expected results: Patients treated with extended-half-life products are expected to report lower treatment burden, higher self-efficacy and better sleep quality, regardless of sociodemographic or clinical factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with a medical diagnosis of hemophilia A or B.
* Patients who, regardless of disease phenotype (mild, moderate or severe), are receiving prophylactic treatment with recombinant or plasma clotting factor concentrates, either short half-life or extended half-life.
* Patients must have maintained the same treatment regimen (SHL or EHL) continuously for at least six months prior to participation.

Exclusion Criteria:

* Patients who have developed inhibitors or antibodies to FVIII or FIX concentrates.
* People with a concomitant diagnosis of other serious or disabling chronic diseases (neurological, oncological, severe psychiatric or rheumatological) that may interfere with the perceived burden of treatment, sleep quality, functionality or perception of self-efficacy.
* Patients with cognitive, linguistic or sensory impairments that prevent them from correctly understanding and completing the questionnaires.
* Patients who are participating in clinical trials or intensive monitoring programmes that may alter their perception of the treatment and generate biases in the evaluation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemophilia A or B, undergoing prophylactic treatment with clotting factor concentrates.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2025-09-13 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of treatment burden at the time of the study. | Screening visit.
  Treatment burden will be assessed using the Spanish version of the Treatment Burden Questionnaire (TBQ). This self-administered multidimensional instrument consists of 15 items that measure the perceived burden of treatment in dimensions such as time spent, emotional impact, physical effort, medical coordination, and interference with daily life. Each item is scored on a Likert scale from 0 (no burden) to 10 (extreme burden). A total score is obtained, with higher values indicating greater perceived burden. This version has demonstrated good internal reliability in the Spanish chronic population (Cronbach's α = 0.89).

SECONDARY OUTCOMES:
Assessment of perceived self-efficacy in health at the time of the study. | Screening visit.
  Perceived self-efficacy in health will be measured using the Spanish version of the General Self-Efficacy Scale (GSE). This questionnaire consists of 10 items with a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree). It assesses the individual's general belief in their ability to cope with difficulties and manage their health. The total score ranges from 10 to 40, with higher values indicating greater self-efficacy. The scale has shown good internal consistency (Cronbach's α = 0.87) in the Spanish population.
Assessment of adherence to treatment at the time of the study. | Screening visit.
  Adherence to treatment will be assessed using the Torres scale. This structured self-report, specific for patients with hemophilia, includes 25 items, grouped into 5 dimensions: awareness of the disease, knowledge of sequelae, treatment difficulties, doctor-patient relationship, and treatment of bleeding episodes. This scale has proven to be valid and reliable for assessing adherence in these patients, with good internal consistency across all dimensions. The total score ranges from 0 to 100, with higher values indicating poorer adherence.
Assessment of sleep quality at the time of the study. | Screening visit.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) in its validated Spanish version. This self-administered questionnaire assesses sleep quality over the last month through 19 items grouped into seven components (latency, duration, efficiency, disturbances, medication use, daytime dysfunction, and subjective sleep quality). Each component is scored from 0 to 3, generating an overall score from 0 to 21, where a score >5 indicates poor sleep quality. Its test-retest reliability and internal consistency have been adequate (Cronbach's α = 0.81).
Assessment of health locus of control at the time of the study. | Screening visit.
  Health locus of control will be measured using the Spanish version of the Multidimensional Health Locus of Control Form C (MHLC-C). This scale consists of 18 items that assess the extent to which people attribute control of their health to internal, medical or random factors. It consists of three subscales of 6 items each, scored on a scale from 1 (total disagreement) to 6 (total agreement). Each subscale generates an independent score. Validation in Spanish has shown good internal reliability (Cronbach's α > 0.70 in all three dimensions).
Assessment of the sociodemographic variable age at the time of the study. | Screening visit.
  The sociodemographic variable age will be assessed by calculating the age (in months) from the date of birth to the date of assessment.
Assessment of the clinical variable number of weekly infusions of clotting factor concentrates at the time of the study. | Screening visit.
  The clinical variable number of weekly infusions of clotting factor concentrates will be assessed by calculating the age (in months) from the date of birth to the date of assessment.

OTHER OUTCOMES:
Assessment of the sociodemographic variable educational level at the time of the study. | Screening visit.
  The sociodemographic variable educational level will be assessed using closed-ended questions (primary education / secondary education / university education / postgraduate education).
Assessment of the sociodemographic variable 'living arrangements at the time of the study'. | Screening visit.
  The sociodemographic variable 'living arrangements' will be assessed using a qualitative variable with three response options: alone / with family / with partner.
Assessment of the clinical variable cohabitation at the time of the study. | Screening visit.
  The clinical variable type of hospital where treatment is received will be a dichotomous variable, with two response options: national referral hospital-CESUR / regional referral hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No